CLINICAL TRIAL: NCT05339906
Title: Study of the Effect of the Auditory Stimulation on Stuttering Symptoms in Patients With a Deficit of Spectral Power in the EEG Beta Frequency Band
Acronym: ZOV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oles Honchar Dnipro National University (Other)
Collaborators: SynthezAI Corp. (Unknown)
Responsible Party: Principal Investigator, Dmytro Chernetchenko, PhD, Associate Professor, Oles Honchar Dnipro National University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ZOV01
Record Dates: First submitted 2022-03-31; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Stuttering, Adult; Stammering
Keywords: Speech disorders; Binaural beats; Auditory stimulation; Stuttering; Stammering
MeSH Terms: conditions — Stuttering; Speech Disorders

STUDY DESIGN:
Intervention Model Description: Audio intervention with the same stimulus for participants with and without stuttering
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZOV.ai digital therapy candidate (Experimental): The arm will use a novel auditory neuro modulating technology that leverages euphonic music tracks with broad-spectrum binaural beats to induce selective EEG spectral power changes to improve stuttering symptoms.
  The total length of the audio stimuli is 5 minutes.
  Interventions: Device: ZOV.ai digital therapy candidate

INTERVENTIONS:
Device: ZOV.ai digital therapy candidate — ZOV.ai is a novel auditory neuro modulating technology that leverages euphonic music tracks with broad-spectrum binaural beats to induce selective EEG spectral power changes to improve stuttering symptoms

SUMMARY:
In this study, the investigators will research the efficacy of a novel auditory neuro modulating technology that leverages euphonic music tracks with broad-spectrum binaural beats to induce selective EEG spectral power changes.

DETAILED DESCRIPTION:
Stuttering is a speech disorder that affects more than 70 million people worldwide, limiting their ability to communicate and socialize. During recent decades, several studies have demonstrated a link between stuttering and a deficit of β EEG spectral power.

In this study, the investigators will research the efficacy of a novel auditory neuro modulating technology that leverages euphonic music tracks with broad-spectrum binaural beats to induce selective EEG spectral power changes. Participants are adults with stuttering and without speech disfluencies from the control group will expose to euphonic binaural stimuli for 5 minutes. The brain electrical activity patterns (EEG) and ECG bio-signals will record prior to, during, and after exposure.

ELIGIBILITY:
Inclusion Criteria:

* Adults with stuttering (stammering) symptoms;

Exclusion Criteria:

* Hearing disabilities;
* Applying other drugs or devices simultaneously;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Speech disfluencies | The outcome measure will be assessed between 5-minute intervals before stimulation, just after and 10 minutes after stimulation
  The total number of repetitions, blocks and prolongations during the speech (assessed by speech therapist) measured before, just after and 10 minutes after auditory stimulation

SECONDARY OUTCOMES:
Heart Rate Variability Stress Index [a.u.] | The outcome measure will be assessed between 5-minute intervals before stimulation, just after and 10 minutes after stimulation
  Stress Level changes assessed by ECG HRV measurements before, just after and 10 minutes after auditory stimulation
Heart Rate Variability meanRR [ms] | The outcome measure will be assessed between 5-minute intervals before stimulation, just after and 10 minutes after stimulation
  Average of RR-intervals array assessed by ECG HRV measurements before, just after and 10 minutes after auditory stimulation
Heart Rate Variability Total Power [ms^2] | The outcome measure will be assessed between 5-minute intervals before stimulation, just after and 10 minutes after stimulation
  Total Power of RR-intervals array spectrogram assessed by ECG HRV measurements before, just after and 10 minutes after auditory stimulation
Heart Rate Variability SDNN [ms] | The outcome measure will be assessed between 5-minute intervals before stimulation, just after and 10 minutes after stimulation
  SDNN value of RR-intervals array assessed by ECG HRV measurements before, just after and 10 minutes after auditory stimulation
Heart Rate Variability RMSSD [ms] | The outcome measure will be assessed between 5-minute intervals before stimulation, just after and 10 minutes after stimulation
  RMSSD value of RR-intervals array assessed by ECG HRV measurements before, just after and 10 minutes after auditory stimulation
EEG spectral power in beta frequency range, [uV^2] | The outcome measure will be assessed between 5-minute intervals before stimulation, just after and 10 minutes after stimulation
  Electrical spectral density in beta frequency range of brain activity measured before, just after and 10 minutes after auditory stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Dmytro Lituiev, PhD, Study Chair — SynthezAI Corp.
Locations (1):
- Oles Honchar Dnipro National University, Dnipro, Dnipropetrovska, Ukraine